CLINICAL TRIAL: NCT03129334
Title: Preventing Prescription Drug Abuse in Middle School Students
Acronym: MSPDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Health Promotion Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Kenneth W Griffin, Senior Research Scientiest, National Health Promotion Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44DA040358-01 (NIH)
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Prescription Drug Abuse (Not Dependent); Substance Use; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LST Middle School Online (Experimental): Students will participate in a series of e-learning modules plus classroom sessions related to drug abuse prevention, including prescription drug abuse
  Interventions: Behavioral: LST Middle School Online
- Treatment as Usual (Control) (No Intervention): Students will not participate in the e-learning modules. They will receive any standard classroom instruction on drug abuse/health education.

INTERVENTIONS:
Behavioral: LST Middle School Online — The adapted intervention will (1) utilize both online e-learning module (self-guided) and classroom-based sessions (facilitator led) to address PDA and concurrent ATOD abuse; (2) positively change social norms and challenge positive expectancies regarding PDA and ATOD abuse; (3) discourage diversion of prescription medications; (4) enhance protective factors by building social and self-regulation skills through interactive learning and behavioral rehearsal scenarios; and (5) incorporate booster sessions.
  Arms: LST Middle School Online

SUMMARY:
This project is designed to test a primary prevention approach to the problem of prescription drug misuse and abuse (PDA) among middle school students. The intervention uses both online e-learning and small group facilitator-led intervention modalities. Middle schools will be randomized to receive the intervention or serve as controls.

DETAILED DESCRIPTION:
While there are a number of drug abuse prevention programs for middle school age youth, relatively few programs focus on preventing prescription drug abuse. Furthermore, due to growing constraints on classroom time, new evidence-based prevention programs are needed that flexibly incorporate the use of online digital technology and classroom/small-group components. The present study is developing and testing an adaptation of the evidence-based substance abuse and violence prevention approach called Life Skills Training (LST). The proposed preventive intervention for middle school PDA will (1) utilize both online digital and face-to-face intervention modalities to address PDA and concurrent ATOD use; (2) positively change social norms and challenge positive expectancies regarding PDA and ATOD use; (3) discourage diversion of prescription medications; and (4) enhance protective factors by building social and self-regulation skills through interactive learning and behavioral rehearsal scenarios. Middle schools will be randomized into either an intervention group that will receive the new intervention or a treatment-as-usual control group that will receive existing health education programming. At the end of the intervention period, and at a 12-month follow-up assessments, we will compare both groups with respect to changes in behaviors, norms, attitudes, and knowledge regarding PDA and substance use.

ELIGIBILITY:
Inclusion Criteria:

* Middle school aged-youth

Exclusion Criteria:

* Significant cognitive impairment or severe learning disabilities, as screened by field staff at participating sites

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4500 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in any prescription drug use in the past year | Post-test (within 2 weeks of completing final session/module of the intervention), 6-month followup, 12-month followup
  The investigators will assess (via questionnaire) key study variables regarding prescription drug abuse and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group at a post-test assessment and 6- and 12-month follow-up assessments.

IPD SHARING:
Plan to Share IPD: No